CLINICAL TRIAL: NCT07042594
Title: A Randomized, Single-blind, Placebo-Controlled Phase I Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses of Subcutaneously Administered RBD1119 in Healthy Participants
Brief Title: Single Ascending Doses Phase I Study to Evaluate the Safety and Pharmacokinetics of RBD1119 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Ribo Life Science Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RBFI2101
Record Dates: First submitted 2025-06-13; First posted 2025-06-29 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RBD1119 SAD experimental group (Experimental): Subjects in SAD experimental groups will receive a single subcutaneous injection of RBD1119 on Day 1.
  Interventions: Drug: RBD1119
- Placebo SAD group (Placebo Comparator): Subjects in SAD placebo groups will receive a single subcutaneous injection of placebo on Day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RBD1119 — Subcutaneously Administered RBD1119 in Healthy Subjects.
  Arms: RBD1119 SAD experimental group
Drug: Placebo — Subcutaneously Administered Placebo in Healthy Subject.
  Arms: Placebo SAD group

SUMMARY:
This is a Randomized, Single-blind, Placebo-Controlled Phase I Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses of Subcutaneously Administered RBD1119 in Healthy Participants.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female healthy participants (non-childbearing potential only), aged 18 to 65 years at screening, inclusive.
* Body mass index (BMI) between 18 and 32 kg/m2, inclusive
* APTT, Prothrombin time (PT), INR, thrombin time (TT) within normal reference range (as per the local laboratory).
* Haematology results within normal range, unless deemed not clinically significant by the Principal Investigator or delegate. Platelet count however must be within normal range per the local laboratory reference ranges.
* Healthy as determined by no clinically significant findings by the Principal Investigator or delegate in medical history, vital signs, physical examination, clinical laboratory assessments, and 12-lead electrocardiogram (ECG).

Main Exclusion Criteria:

* Any uncontrolled or serious disease that may interfere with participation in the clinical trial and/or put the participant at significant risk (according to Principal Investigator or delegate's judgment) if he/she participates in the clinical trial.
* History or presence of cardiovascular disease (including peripheral artery and cerebrovascular disease).
* Systolic blood pressure (SBP) is less than 90 or greater than 140 mmHg and/or diastolic blood pressure (DBP) is less than 50 or greater than 95 mmHg after 10 minutes of supine rest, unless determined by the Principal Investigator or delegate to be not clinically significant.
* Diagnosis of diabetes mellitus, history of gestational diabetes that has not been fully resolved is not permitted.
* History or presence of:

  * Bleeding disorder(s) and/or at risk of bleeding, including relevant familial history, such as Hemophilia A, Hemophilia B, Wiskott-Aldrich syndrome, von Willebrand disease (vWD);
  * Clinically significant anemia, in the opinion of the Principal Investigator or delegate;
  * Thromboembolic diseases;
  * Bleeding in the gastrointestinal tract or central nervous system;
  * Anticipated need for oral surgery or tooth extractions during the trial period;
  * Bleeding in the genitourinary tract;
  * Gum disease or active gum bleeding;
  * Planned surgery during the trial period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v5.0 | Up to Day 85

SECONDARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v5.0 | After day 85
To characterize the pharmacokinetics (PK) as maximum plasma concentration (Cmax) of RBD1119 in healthy participants | Up to 48 hours post-dose
To evaluate the pharmacodynamics (PD) effect of RBD1119 as percentage change from baseline in intrinsic coagulation pathway related antigen levels in healthy participants. | Up to Day 169.
To characterize the pharmacokinetics (PK) as Time to reach Cmax (Tmax) of RBD1119 in healthy participants | Up to 48 hours post-dose
To characterize the pharmacokinetics (PK) as area under the plasma concentration-time curve from the time zero to the last measurable concentration (AUC0-t) of RBD1119 in healthy participants | Up to 48 hours post-dose
To characterize the pharmacokinetics (PK) as area under the plasma concentration-time from time zero to infinity (AUC0-inf) of RBD1119 in healthy participants | Up to 48 hours post-dose
To characterize the pharmacokinetics (PK) as apparent terminal elimination half-life (t1/2) of RBD1119 in healthy participants | Up to 48 hours post-dose
To evaluate the pharmacodynamics (PD) effect of RBD1119 as percentage change from baseline in intrinsic coagulation pathway related activity levels in healthy participants. | Up to Day 169.
To evaluate the pharmacodynamics (PD) effect of RBD1119 as percentage change from baseline in APTT in healthy participants. | Up to Day 169.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Gabrielsen, MD, Study Chair — Suzhou Ribo Life Science Co. Ltd.
Locations (1):
- CMAX Clinical Research, Adelaide, Australia